CLINICAL TRIAL: NCT06459882
Title: Effect of Progressive Relaxation Exercises on Dyspnea and Comfort Level in Individuals With Chronıc Obstructive Lung Disease: A Randomized Controlled Study
Brief Title: Effect of Progressive Relaxation Exercıses on Dyspnea and Comfort Level in Individuals With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Aysegul Celik, Asst. Prof., RN, MSc, PhD, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BakircaU
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Copd; Dyspnea; Nursing Caries
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive relaxation exercises (Experimental): Patients in the intervention group received 30-minute progressive relaxation exercises for 6 weeks.
  Interventions: Behavioral: progressive relaxation exercises
- control (No Intervention): Patients in the control group did not receive any intervention other than standard care practices.

INTERVENTIONS:
Behavioral: progressive relaxation exercises — Patients in the intervention group received 30-minute progressive relaxation exercises for 6 weeks
  Arms: progressive relaxation exercises

SUMMARY:
The study is a randomised controlled experimental study conducted to examine the effect of progressive relaxation exercises on dyspnea and comfort level in individuals with chronic obstructive pulmonary disease. The study was conducted between January and August 2023 in the Internal Medicine Clinic of Izmir Urla State Hospital. Stratified and block randomisation method was used in the study and 42 patients, 21 intervention group and 21 control group, were completed. Patients in the intervention group received 30-minute progressive relaxation exercises for 6 weeks. Patients in the control group did not receive any intervention other than standard care practices. The data of the study were collected by face-to-face interview method using the Descriptive Information Form, Medical Research Council Dyspnea Scale, General Comfort Scale-Short Form and Patient Follow-up Form. Descriptive statistics, Shapiro Wilk test, Levene's test, Mauchly's W test, independent sample T test, Mann Whitney U test, dependent sample t test, Wilcoxon Signed Ranks test, Friedman test, Benferoni test and Fisher's Exact test were used to analyse the data obtained from the study. It was determined that the mean dyspnea level scores of the patients in the intervention group at week 6 were lower than the control group and this difference between the groups was statistically significant (p<0.05). It was determined that the decrease in the mean comfort level scores of the patients in the intervention group according to the follow-up periods was statistically significant (p<0.05). According to the results of the study, progressive relaxation exercises can be recommended as an effective nursing intervention to provide dyspnea management in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* Inpatient treatment in the Internal Medicine Clinic of Izmir Urla State Hospital
* Standardised Mini Mental Test score ≥24
* Dyspnea severity ≥2 according to the MMRC dyspnoea scale
* Diagnosed with Stage II and Stage III COPD according to GOLD criteria
* Functional competence to participate in progressive relaxation exercises
* Able to access and use a smartphone
* COPD patients who agreed to participate in the study.

Exclusion Criteria:

* Have any speech and hearing problems
* Lung disease other than COPD, physical dependence and psychiatric illness diagnosed with
* COPD patients in the acute exacerbation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
dyspnea level | baseline, week 3, and week 6
  Medical Research Council Scale: MMRC is an easily applicable 5-item scale that shows similar results with lung function tests and arterial blood gas measurement and is recommended for use in determining the dyspnea levels of COPD patients in GOLD guidelines. The dyspnea level is graded between 0-4. A score of 0 indicates the absence of dyspnea, and an increase in the rating indicates an increase in the severity of dyspnea.
comfort level | baseline, week 3, and week 6
  The scale consists of 28 items and three sub-dimensions: relief (9 items), relaxation (9 items) and overcoming problems (10 items). The lowest value of 1 indicates a low comfort level and the highest value of 6 indicates a high comfort level. In this study, the Cronbach alpha reliability coefficient of the scale was 0.74 for the intervention group and 0.82 for the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Çelik, PhD, Principal Investigator — Izmir Bakircay University
Locations (1):
- Izmir Bakırcay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No